CLINICAL TRIAL: NCT06610279
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, 3-Part Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-951 in Healthy Subjects
Brief Title: A Study of TAK-951 in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on the Sponsor's decision attributed to the benefit-risk profile derived from the Part 1 data of this study.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-951-1008
Record Dates: First submitted 2024-09-21; First posted 2024-09-24 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteers
Keywords: TAK-951

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Pooled Placebo (Placebo Comparator): Participants will receive a single SC dose of TAK-951 matching placebo on Day 1.
  Interventions: Drug: Placebo
- Part 1, Cohort 1: TAK-951 Dose 1 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 1 on Day 1.
  Interventions: Drug: TAK-951
- Part 1, Cohort 2: TAK-951 Dose 2 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 2 on Day 1.
  Interventions: Drug: TAK-951
- Part 1, Cohort 3: TAK-951 Dose 3 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 3 on Day 1.
  Interventions: Drug: TAK-951
- Part 1, Cohort 4: TAK-951 Dose 4 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 4 on Day 1.
  Interventions: Drug: TAK-951
- Part 1, Cohort 5: TAK-951 Dose 5 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 5 on Day 1.
  Interventions: Drug: TAK-951
- Part 1, Cohort 6: TAK-951 Dose 6 (Experimental): Participants will receive a single SC dose of TAK-951 Dose 6 on Day 1.
  Interventions: Drug: TAK-951
- Part 2: TAK-951 Multiple Rising Doses (Experimental): Participants will receive multiple rising SC doses of TAK-951 twice daily (BID) or 3 times a day (TID) in Part 2.
  Interventions: Drug: TAK-951
- Part 3: TAK-951 Multiple Dose Titration (Experimental): Participants will receive multiple rising SC doses of TAK-951 once daily (QD), BID, or TID from Days 1 to 5 followed by a washout period of 2 to 7 days and a single redose on any day from Days 8 to 13 in Part 3.
  Interventions: Drug: TAK-951

INTERVENTIONS:
Drug: TAK-951 — TAK-951 SC injection
  Arms: Part 1, Cohort 1: TAK-951 Dose 1; Part 1, Cohort 2: TAK-951 Dose 2; Part 1, Cohort 3: TAK-951 Dose 3; Part 1, Cohort 4: TAK-951 Dose 4; Part 1, Cohort 5: TAK-951 Dose 5; Part 1, Cohort 6: TAK-951 Dose 6; Part 2: TAK-951 Multiple Rising Doses; Part 3: TAK-951 Multiple Dose Titration
Drug: Placebo — TAK-951 matching placebo SC injection
  Arms: Part 1: Pooled Placebo

SUMMARY:
Feeling sick in the stomach (nausea) or throwing up (vomiting) are among the most common symptoms during treatment with medicines. It is hoped that a medicine called TAK-951 may help people to not feel sick in the stomach or throw up. The main aim of this study is to learn about side effects of TAK-951 when given as a single or multiple doses to healthy adults. Side effects are medical problems thought to be caused by the study treatment. Another aim is to learn how a healthy adult's body processes TAK-951 (this is called pharmacokinetics or PK). In this study, participants will receive either TAK-951 or placebo. The placebo looks like TAK-951 but does not have any medicine in it. Both TAK-951 and placebo will be given as an injection directly under the skin. This is called subcutaneous or subcutaneous (SC).

The study will be conducted in 3 parts:

* In Part 1, participants will be given one SC injection of either TAK-951 or placebo.
* In Part 2, participants will receive up to three daily SC injections of either TAK-951 or placebo of the same dose
* In Part 3, participants will receive one SC injection of either TAK-951 or placebo and another SC injection up to 1 week later.

Participants will be checked for their health either 28 days after the last injection (Parts 1 and 2) or 14 days after the last injection (Part 3).

ELIGIBILITY:
Inclusion Criteria

To be eligible for participation in this study, the participant must:

1. Understand the study procedures and agree to participate by providing written informed consent.
2. Be willing and able to comply with all study procedures and restrictions.
3. Be a healthy man or woman aged 18 to 55 years, inclusive, at the screening visit.
4. Be a continuous nonsmoker who has not used nicotine and tobacco-containing products for at least 3 months prior to dosing and throughout the study.
5. Have a body mass index (BMI) greater than equal to (≥)18 and less than equal to (≤)32 kilograms per meter square (kg/m^2) at the screening visit.
6. Be judged to be in good health (e.g., no evidence of psychiatric, hepatic, renal, pulmonary, or cardiovascular (CV) disease) by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, ECG, and vital sign measurements performed at the screening visit and before administration of the initial dose of study drug or invasive procedure.
7. Meet the following birth control requirements:

   * Is a male participant who is sterile or agrees to use an appropriate method of contraception, including a condom with or without spermicidal cream or jelly, from the first dose of study drug until 30 days after the last dose of study drug. No restrictions are required for a vasectomized male participant provided the participant is at least 1 year after bilateral vasectomy procedure before the first dose of study drug. A male participant whose vasectomy procedure was performed less than 1 year before the first dose of study drug must follow the same restrictions as a non-vasectomized man. Appropriate documentation of surgical procedure should be provided.
   * Is a male participant who agrees not to donate sperm from the first dose of study drug until 30 days after the last dose of study drug.
   * Women of childbearing potential are eligible for the study provided they have a negative pregnancy test, are not lactating or breastfeeding, and are willing and agreeable to use highly effective contraception during the study and up to 30 days after the last dose of study drug.
   * Is a female participant of nonchildbearing potential, defined by at least 1 of the following criteria:

     1. Postmenopausal (defined as 12 months of spontaneous amenorrhea in females aged greater than (>)45 years or 6 months of spontaneous amenorrhea in females aged >45 years with serum follicle-stimulating hormone (FSH) levels >40 milli-international units per milliliter [mIU/mL]). Appropriate documentation of FSH levels is required.
     2. Surgically sterile by hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
     3. Had a bilateral tubal ligation with appropriate documentation of surgical procedure.
     4. Has a congenital condition resulting in no uterus. Exclusion Criteria

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. The participant has participated in another investigational study within 4 weeks (or based on local regulations) or within 5 half-lives, whichever is longest, of the investigational product before the screening visit. The 4-week or 5 half-lives window will be derived from the date of the last dose and/or AE related to the study procedure in the previous study to the screening visit of the current study.
2. The participant is an employee of the sponsor or study site or immediate family member (e.g., spouse, parent, child, sibling) of the sponsor or study site.
3. The participant has a history of significant multiple and/or severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food, as determined by the investigator.
4. The participant has a known hypersensitivity or contraindication to any component of TAK-951.
5. The participant has a positive pregnancy test or is lactating or breastfeeding.
6. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency antibody/antigen, at the screening visit.
7. The participant had major surgery or donated or lost 1 unit of blood (approximately 500 milliliters [mL]) within 4 weeks before the screening visit.
8. The participant is unable to refrain from or anticipates using any medications including herbal medicines beginning approximately 7 days before administration of the first dose of study drug, throughout the study until 2 days after discharge.
9. The participant is unable to refrain from or anticipates using marijuana or cannabis-containing products beginning approximately 7 days before administration of the first dose of study drug, throughout the study until after the last pharmacokinetic (PK) dose.
10. The participant has a history or presence of alcoholism or drug abuse within the past 2 years prior to dosing, or frequent or heavy use (i.e., near-daily) of medical or recreational cannabis in the past 3 months before screening, as determined by the investigator.
11. The participant drinks alcohol in excess of 7 drinks/week for women or 14 drinks/week for men (where 1 drink=5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor [45% alcohol]) within 3 months before screening.
12. The participant has a positive alcohol test or urine drug screen results at screening or check-in.
13. The participant has had a previous major psychiatric disorder.
14. The participant has a history or presence of:

    * 3 or more incidences of vasovagal syncope within the last 5 years prior to screening; or
    * A family history of unexplained sudden death or channelopathy; or
    * Brugada syndrome (i.e., right bundle branch block [RBBB] pattern with ST-elevation in leads V1-V3); or
    * Cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, sick sinus syndrome, pulmonary congestion, symptomatic or significant cardiac arrhythmia, second-degree atrioventricular (AV) block type 2, third-degree AV block, prolonged QT interval with Fridericia correction method (QTcF) interval, hypokalemia, hypomagnesemia, or conduction abnormalities; or
    * Risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome); or
    * Any clinically significant ECG findings or medical history including: long or short QTcF (over 450 milliseconds (msec) or less than 360 msec), bifascicular block or QRS ≥120 msec or PR interval >210 msec at screening or Day 1 pre-Hour 0; or
    * The participant has a documented history of sinus bradycardia (<45 beats per minute [bpm]), sinoatrial block or sinus pause ≥3 seconds.
15. The participant has an average semirecumbent blood pressure (BP) less than (<)90/60 millimeters of mercury (mm Hg) or >140/90 mm Hg from screening to predose, inclusive. Any assessments on Day -1 that do not meet this criterion must be discussed with the medical monitor for approval.
16. The participant has an average semirecumbent heart rate (HR) (pulse) <55 or >100 bpm at any time point from screening to predose, inclusive. Participants with an average HR (pulse) <55 bpm can be enrolled only with medical monitor approval. Any assessments after admission with an average HR (pulse) <55 bpm at any time point, from Day -2 to predose (inclusive), will be left to the judgment of the investigator, unless HR (pulse) is <50 bpm, which must be discussed with the medical monitor for approval.
17. The participant has orthostatic hypotension defined as a decrease in systolic blood pressure (SBP) ≥20 mm Hg or a decrease in diastolic blood pressure (DBP) ≥10 mm Hg at approximately 3 minutes of standing when compared with BP from the semirecumbent position at screening to predose assessments, inclusive. In asymptomatic participants, any assessments after screening that do not meet this criterion may be repeated after the participant has remained in the semirecumbent or supine position for 15 minutes. If the repeat assessment is exclusionary based on the above criterion, the participant will not be eligible. If the repeat assessment is not exclusionary, the participant will be eligible.
18. The participant has postural orthostatic tachycardia, defined as an increase of >30 bpm or pulse >120 bpm at approximately 3 minutes of standing, at screening to predose assessments, inclusive. Any assessments after screening that do not meet this criterion may be repeated with the participant remaining standing for up to a total of 5 minutes, provided that the participant remains asymptomatic. If the repeat assessment occurring within 5 minutes is exclusionary based on the above criterion, the participant will not be eligible. A confirmed orthostatic increase of >30 bpm, but <40 bpm, on 1 or more Day -1 assessments may not be considered exclusionary if not considered clinically significant by the investigator and the medical monitor. Such assessments must be discussed with the medical monitor before determination that the participant is eligible to proceed.
19. The participant has a known or suspected current coronavirus disease 2019 (COVID-19) infection or is at risk of COVID-19 infection as assessed by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ICON, Lenexa, Kansas
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 7 January 2022 to 21 September 2023.
Pre-assignment Details: A total of 48 healthy participants were enrolled in Part 1 Single Rising Dose (SRD) of the study and randomized to receive either placebo or TAK-951. This study was terminated after completion of Part 1 following the Sponsor's decision attributed to the benefit-risk profile derived from the Part 1 data. Hence, no participants were enrolled in Parts 2 and 3.
Groups:
- Part 1: Pooled Placebo: Participants received a single subcutaneous (SC) dose of TAK-951 matching placebo on Day 1.
- Part 1, Cohort 1: TAK-951 Dose 1: Participants received a single SC dose of TAK-951 Dose 1 on Day 1.
- Part 1, Cohort 2: TAK-951 Dose 2: Participants received a single SC dose of TAK-951 Dose 2 on Day 1.
- Part 1, Cohort 3: TAK-951 Dose 3: Participants received a single SC dose of TAK-951 Dose 3 on Day 1.
- Part 1, Cohort 4: TAK-951 Dose 4: Participants received a single SC dose of TAK-951 Dose 4 on Day 1.
- Part 1, Cohort 5: TAK-951 Dose 5: Participants received a single SC dose of TAK-951 Dose 5 on Day 1.
- Part 1, Cohort 6: TAK-951 Dose 6: Participants received a single SC dose of TAK-951 Dose 6 on Day 1.
- Part 2, TAK-951 Multiple Rising Dose Cohort: Participants were planned to receive multiple rising SC doses of TAK-951 twice daily (BID) or 3 times a day (TID) in Part 2.
- Part 3, TAK-951 Multiple Dose Titration Cohort: Participants were planned to receive multiple rising SC doses of TAK-951 once daily (QD), BID, or TID from Days 1 to 5 followed by a washout period of 2 to 7 days and a single redose on any day from Days 8 to 13 in Part 3.
Period: Part 1
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6 | Part 2, TAK-951 Multiple Rising Dose Cohort | Part 3, TAK-951 Multiple Dose Titration Cohort
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6 | Part 2, TAK-951 Multiple Rising Dose Cohort | Part 3, TAK-951 Multiple Dose Titration Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6 | Part 2, TAK-951 Multiple Rising Dose Cohort | Part 3, TAK-951 Multiple Dose Titration Cohort
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study treatment. This study was terminated after completion of Part 1 following the Sponsor's decision attributed to the benefit-risk profile derived from the Part 1 data. Hence, no participants were enrolled in Parts 2 and 3.
Groups:
- Part 1: Pooled Placebo: Participants received a single SC dose of TAK-951 matching placebo on Day 1.
- Part 2, TAK-951 Multiple Rising Dose Cohort: Participants were planned to receive multiple rising SC doses of TAK-951 BID or TID in Part 2.
- Part 3, TAK-951 Multiple Dose Titration Cohort: Participants were planned to receive multiple rising SC doses of TAK-951 QD, BID, or TID from Days 1 to 5 followed by a washout period of 2 to 7 days and a single redose on any day from Days 8 to 13 in Part 3.
- Total: Total of all reporting groups
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6 | Part 2, TAK-951 Multiple Rising Dose Cohort | Part 3, TAK-951 Multiple Dose Titration Cohort | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.36 (10.68) | 34.5 (10.07) | 35.2 (5.91) | 31.7 (9.71) | 30.0 (8.92) | 28.0 (11.10) | 40.2 (10.09) |  |  | 33.3 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 2 | 0 | 2 | 3 | 0 | 0 | 10
  Male | 10 | 5 | 6 | 4 | 6 | 4 | 3 | 0 | 0 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 5 | 0 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 13
  Ethnicity: Not Hispanic or Latino | 7 | 6 | 4 | 4 | 5 | 5 | 4 | 0 | 0 | 35
  Ethnicity: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race: Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Race: Black or African American | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 5
  Race: White | 8 | 4 | 3 | 4 | 6 | 5 | 6 | 0 | 0 | 36
  Race: More than one race | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Race: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug. An AE can be any unfavorable and unintended sign (including physical examinations, vital signs, electrocardiogram (ECG), laboratory assessment findings), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug.
Time Frame: From the first dose of study drug up to Day 29 in Part 1
Population: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 6 | 4 | 5 | 6 | 5 | 4 | 6

2. Primary Outcome: Part 2: Number of Participants With TEAEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug. An AE can be any unfavorable and unintended sign (including physical examinations, vital signs, ECG, laboratory assessment findings), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE was defined as an AE that started or worsened after first study drug administration and within 30 days of last dose of study drug.
Time Frame: From the first dose of study drug up to Day 33 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

3. Primary Outcome: Part 3: Number of Participants With TEAEs
Description: as for outcome 2
Time Frame: From the first dose of study drug up to Day 27 in Part 3
Population: Data was not collected as no participants were enrolled in Part 3 due to study termination.
Arm/Group | Part 3, TAK-951 Multiple Dose Titration Cohort
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration of TAK-951
Description: Due to confidentiality reasons and chances of exposing the doses for TAK-951, the data for this pharmacokinetic outcome measure was not reported.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Part 1: AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours for TAK-951
Description: as for outcome 4
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 1
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Part 1: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-951
Description: as for outcome 4
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Part 1: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration for TAK-951
Description: as for outcome 4
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Part 1: Tmax: Time of First Occurrence of Cmax for TAK-951
Description: as for outcome 4
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Part 1: t1/2z: Terminal Disposition Phase Half-life for TAK-951
Description: as for outcome 4
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Part 1: CL/F: Apparent Clearance After Extravascular Administration of TAK-951
Description: Apparent clearance after extravascular administration was calculated as Dose/AUC∞. Due to confidentiality reasons and chances of exposing the doses for TAK-951, the data for this pharmacokinetic outcome measure was not reported.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Part 1: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration
Description: Apparent volume of distribution during the terminal disposition phase after extravascular administration was calculated as (CL/F)/λz, where λz is the terminal elimination rate constant. Due to confidentiality reasons and chances of exposing the doses for TAK-951, the data for this pharmacokinetic outcome measure was not reported.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 3 in Part 1
Reporting Status: Not Posted

12. Secondary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) for TAK-951 on Day 1 of Drug Dosing
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

13. Secondary Outcome: Part 2: Time of First Occurrence of Cmax (Tmax) for TAK-951 on Day 1 of Drug Dosing
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

14. Secondary Outcome: Part 2: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC24) for TAK-951 on Day 1 of Drug Dosing
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

15. Secondary Outcome: Part 2: AUCτ: Area Under the Plasma Concentration-time Curve During a Dosing Interval for TAK-951 on Day 1
Description: Tau (τ) indicates the length of the dosing interval.
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

16. Secondary Outcome: Part 2: AUCτ for TAK-951 at Steady State
Description: τ indicates the length of the dosing interval.
Time Frame: Predose and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

17. Secondary Outcome: Part 2: AUC24 for TAK-951 at Steady State
Time Frame: Predose on Day 1 and at multiple time points post-dose up to 24 hours on Day 1 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

18. Secondary Outcome: Part 2: Cmax,ss: Maximum Observed Concentration at Steady State for TAK-951
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

19. Secondary Outcome: Part 2: Tmax for TAK-951 at Steady State
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

20. Secondary Outcome: Part 2: Terminal Disposition Phase Half-life (t1/2z) for TAK-951 at Steady State
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

21. Secondary Outcome: Part 2: Apparent Clearance After Extravascular Administration (CL/F) for TAK-951 at Steady State
Description: Apparent clearance after extravascular administration was to be calculated as Dose/AUCτ after multiple dosing.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 2: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration (Vz/F) for TAK-951 at Steady State
Description: Apparent volume of distribution during the terminal disposition phase after extravascular administration was to be calculated as (CL/F)/λz at steady state, with λz as the terminal elimination rate constant.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 2: Ctrough: Observed Plasma Concentration at the End of a Dosing Interval for TAK-951 at Steady State
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

24. Secondary Outcome: Part 2: Rac[AUC]: Accumulation Ratio Based on AUCτ for TAK-951 at Steady State
Description: Rac[AUC] was to be calculated as the ratio of AUCτ at steady state/AUCτ after a single dose.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

25. Secondary Outcome: Part 2: Rac[Cmax]: Accumulation Ratio Based on Cmax for TAK-951 at Steady State
Description: Rac[Cmax] was to be calculated as the ratio of Cmax at steady state/Cmax after a single dose.
Time Frame: Predose on Day 1 and at multiple time points post-dose up to Day 7 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

26. Secondary Outcome: Part 3: Number of Participants With AEs
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug. An AE can be any unfavorable and unintended sign (including physical examinations, vital signs, ECG, laboratory assessment findings), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug.
Time Frame: From the re-treatment dose of study drug (any day from Days 8 to 13) up to Day 27 in Part 3
Population: Data was not collected as no participants were enrolled in Part 3 due to study termination.
Arm/Group | Part 3, TAK-951 Multiple Dose Titration Cohort
Number analyzed (Participants) | 0

27. Secondary Outcome: Part 1: Number of Participants Based on Antidrug Antibodies (ADA) Status in Serum
Description: A 3-tiered ADA testing strategy was used in this study. A sample was initially screened for ADA by the ADA screening assay. Any positive sample in the screening assay was considered a potential positive, which was confirmed for true positivity by the confirmatory assay. If a sample was confirmed as an ADA true positive, ADA titer was assessed. ADA-positive was defined as participants who have confirmed positive ADA status in at least 1 postbaseline assessments. ADA-negative was defined as participants who did not have a confirmed positive ADA status in any postbaseline assessment. For ADA-positive only, high ADA titer was defined as participant who had at least 1 postbaseline ADA titer >16; low ADA titer was defined as participant whose postbaseline ADA titers were all ≤16 and data is presented accordingly for each of these categories.
Time Frame: Predose on Day 1 and post-dose on Days 14 and 29 in Part 1
Population: The Immunogenicity Analysis Set included all participants who received at least 1 dose of study treatment and had the baseline sample and at least 1 postbaseline sample ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Day 1: Negative | 12 | 6 | 6 | 6 | 5 | 6 | 6
  Day 1: Positive: Low Titer | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 1: Positive: High Titer | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: Negative | 12 | 6 | 6 | 6 | 5 | 6 | 6
  Day 14: Positive: Low Titer | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 14: Positive: High Titer | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29: Negative | 12 | 6 | 6 | 6 | 5 | 6 | 6
  Day 29: Positive: Low Titer | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day 29: Positive: High Titer | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Part 2: Number of Participants With ADA
Time Frame: Predose on Day 1 and post-dose on Days 14 and 29 in Part 2
Population: Data was not collected as no participants were enrolled in Part 2 due to study termination.
Arm/Group | Part 2, TAK-951 Multiple Rising Dose Cohort
Number analyzed (Participants) | 0

29. Secondary Outcome: Part 3: Number of Participants With ADA
Time Frame: Predose on Day 1 and post-dose on Days 14 and 29 in Part 3
Population: Data was not collected as no participants were enrolled in Part 3 due to study termination.
Arm/Group | Part 3, TAK-951 Multiple Dose Titration Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to Day 29 in Part 1
Description: The Safety Analysis Set included all participants who were randomized and received at least 1 dose of study treatment was used to collect safety data for Part 1. This study was terminated after completion of Part 1 following the Sponsor's decision attributed to the benefit-risk profile derived from the Part 1 data. Hence, no participants were enrolled in Parts 2 and 3 and no data for the same could be presented.
Arm/Group | Part 1: Pooled Placebo | Part 1, Cohort 1: TAK-951 Dose 1 | Part 1, Cohort 2: TAK-951 Dose 2 | Part 1, Cohort 3: TAK-951 Dose 3 | Part 1, Cohort 4: TAK-951 Dose 4 | Part 1, Cohort 5: TAK-951 Dose 5 | Part 1, Cohort 6: TAK-951 Dose 6
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/12 | 4/6 | 5/6 | 6/6 | 5/6 | 4/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pooled Placebo (N=12) | Part 1, Cohort 1: TAK-951 Dose 1 (N=6) | Part 1, Cohort 2: TAK-951 Dose 2 (N=6) | Part 1, Cohort 3: TAK-951 Dose 3 (N=6) | Part 1, Cohort 4: TAK-951 Dose 4 (N=6) | Part 1, Cohort 5: TAK-951 Dose 5 (N=6) | Part 1, Cohort 6: TAK-951 Dose 6 (N=6)
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pooled Placebo (N=12) | Part 1, Cohort 1: TAK-951 Dose 1 (N=6) | Part 1, Cohort 2: TAK-951 Dose 2 (N=6) | Part 1, Cohort 3: TAK-951 Dose 3 (N=6) | Part 1, Cohort 4: TAK-951 Dose 4 (N=6) | Part 1, Cohort 5: TAK-951 Dose 5 (N=6) | Part 1, Cohort 6: TAK-951 Dose 6 (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 1 | 3 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 2 | 2 | 5 | 2 | 4 | 5
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT06610279/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT06610279/SAP_001.pdf